CLINICAL TRIAL: NCT01507649
Title: The Effect of a Telephone-based Cognitive-behavioral Intervention on Postnatal Depression: a Randomized Controlled Trial
Brief Title: Effect of a Telephone-based Intervention on Postnatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09101031
Record Dates: First submitted 2012-01-03; First posted 2012-01-11 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Postnatal Depression
Keywords: postnatal depression; quality of life
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Telephone-based intervention (Experimental)
  Interventions: Behavioral: telephone-based cognitive-behavioral intervention

INTERVENTIONS:
Behavioral: telephone-based cognitive-behavioral intervention — The intervention is based on the cognitive-behavioral approach. It consists of five, 30-minutes sessions delivered weekly from postpartum week one to week five via telephone.
  Arms: Telephone-based intervention

SUMMARY:
Purpose: To evaluate the effectiveness of a telephone-based intervention using cognitive-behavioral approach in preventing postnatal depression and improving quality of life in first-time Chinese mothers.

Hypothesis: Women who receive the telephone-based cognitive-behavioral intervention will have a lower level of depressive symptoms (primary outcome) and a higher level of quality of life at 6 weeks and 6 months postpartum than those who receive the usual postpartum care.

Design and subjects: Randomized controlled trial is used. A sample of postpartum women with high risk of postnatal depression (EPDS > 9, n = 498) will be randomly assigned to either the experimental (n = 249) or the control groups (n = 249). The experimental group receives the intervention and the control group receives usual postpartum care.

Study instruments: EPDS and Medical Outcomes Study Short Form Health Survey (SF-12).

Interventions: The intervention is based on the cognitive-behavioral approach. It consists of five, 30-minutes sessions delivered weekly from postpartum week one to week five via telephone.

Main outcome measures and analysis: Outcomes on postnatal depression and quality of life will be measured by EPDS and SF-12, respectively, at 6 weeks and 6 months postpartum. A repeated-measures multivariate analysis of variance will be used to compare differences between two groups.

DETAILED DESCRIPTION:
The aim of this study is to design, implement and evaluate a telephone-based intervention using cognitive-behavioral approach for first-time mothers during the immediate postpartum period. The objective is to evaluate the effect of a telephone-based intervention using cognitive-behavioral approach on postnatal depression and quality of life at 6 weeks and 6 months postpartum.

A longitudinal, randomized, pre and post-test control group design will be used. This design involves providing a 5-week telephone-based intervention using cognitive-behavioral approach at the immediate postpartum period (first five weeks postpartum) to women with high risk of postnatal depression. The experimental group receives the intervention on top of the usual postpartum care, while the control group receives the usual postpartum care only. Participants will be recruited through the postnatal wards at three regional public hospitals in Hong Kong. Eligible participants will be randomly assigned to either the telephone-based intervention or control group. The allocation schedule will be prepared in advanced using a restricted randomization scheme (random permutated blocks of six) by a random number table. The random numbers will be placed in sequentially numbered, opaque and sealed envelopes. After the women have given informed written consent at 2-3 days postpartum at the postnatal units, the research assistant will open the envelope containing the group assignment.

Participants will be postpartum women who meet the inclusion and exclusion criteria. The research nurse will determine if the women meet the sample inclusion criteria from their records. Potential eligible participants will be approached on the second or third postpartum day at the postnatal units. Women will be provided with essential information on the nature of the study and invited to complete the EPDS. Women who score above 9 on EPDS are considered at risk of postnatal depression and they will be invited to participate in the study. Verbal and written explanations of the purpose and the procedure of the study will be provided by the research nurse and written consent will be obtained from women who agree to participate in the study. Participants will be asked to complete the baseline measures, including EPDS and SF-12. Post-test measures will be collected at 6 weeks and 6 months postpartum through mail.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above
* first-time mother
* have given birth to a single full-term healthy baby
* able to speak and read the Chinese language
* Hong Kong residents
* score above 9 on EPDS.

Exclusion Criteria:

* single
* having complications after delivery
* having regular follow up with psychiatrists
* currently taking antidepressant or antipsychotic drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | 6 weeks and 6 months postpartum
  change from baseline depressive symptoms at 6 weeks postpartum and change from baseline depressive symptoms at 6 months postpartum

SECONDARY OUTCOMES:
Change in quality of life | 6 weeks and 6 months postpartum
  change from baseline quality of life at 6 weeks postpartum and change from baseline quality of life at 6 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ngai FW, Wong PW, Chung KF, Leung KY. The effect of a telephone-based cognitive behavioral therapy on quality of life: a randomized controlled trial. Arch Womens Ment Health. 2017 Jun;20(3):421-426. doi: 10.1007/s00737-017-0722-0. Epub 2017 Mar 30. PMID 28361441
- [Derived] Ngai FW, Wong PW, Chung KF, Leung KY. The effect of telephone-based cognitive-behavioural therapy on parenting stress: A randomised controlled trial. J Psychosom Res. 2016 Jul;86:34-8. doi: 10.1016/j.jpsychores.2016.03.016. Epub 2016 Apr 16. PMID 27302544